CLINICAL TRIAL: NCT04425902
Title: Effects of GSK3640254 on the Single-Dose Pharmacokinetics of Probe Substrates (Caffeine, Metoprolol, Montelukast, Flurbiprofen, Omeprazole, Midazolam, Digoxin, and Pravastatin) in Healthy Subjects
Brief Title: Evaluation of Pharmacokinetic Interaction Between GSK3640254 and Caffeine, Metoprolol, Montelukast, Flurbiprofen, Omeprazole, Midazolam, Digoxin, and Pravastatin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213052
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Results first posted 2022-05-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
Keywords: GSK3640254; Human immunodeficiency virus (HIV) infections; Drug interaction; Pharmacokinetics; Probe substrate
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Infections | interventions — GSK3640254; Caffeine; Metoprolol; montelukast; Flurbiprofen; Omeprazole; Midazolam; Digoxin; Pravastatin

STUDY DESIGN:
Intervention Model Description: This is a single-sequence, one-way drug interaction study.
Masking Description: This is a single-group, single-arm study that has no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Probe Substrates/GSK3640254 200 mg/Probe Substrates+GSK3640254 (Experimental): All participants will receive a single dose of treatment A: Probe substrates (caffeine 200 milligram [mg], metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) on Day 1; followed by treatment B- GSK3640254 200 mg on Days 11 to 20; further followed by treatment C: Probe substrates (Caffeine 200 mg, metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) co-administered with GSK3640254 200 mg on Day 21.
  Interventions: Drug: GSK3640254 200 mg; Drug: Caffeine 200 mg; Drug: Metoprolol 100 mg; Drug: Montelukast 10 mg; Drug: Flurbiprofen 100 mg; Drug: Omeprazole 40 mg; Drug: Midazolam 5 mg (2.5 mL); Drug: Digoxin 0.25 mg; Drug: Pravastatin 40 mg

INTERVENTIONS:
Drug: GSK3640254 200 mg — GSK3640254 will be available as oral tablets at unit dose strength of 100 mg.
Drug: Caffeine 200 mg — Caffeine will be available as oral tablets at unit dose strength of 200 mg.
Drug: Metoprolol 100 mg — Metoprolol will be available as oral tablets at unit dose strength of 100 mg.
Drug: Montelukast 10 mg — Montelukast will be available as oral tablets at unit dose strength of 10 mg.
Drug: Flurbiprofen 100 mg — Flurbiprofen will be available as oral tablets at unit dose strength of 100 mg.
Drug: Omeprazole 40 mg — Omeprazole will be available as oral capsules at unit dose strength of 40 mg.
Drug: Midazolam 5 mg (2.5 mL) — Midazolam will be available as syrup for oral administration at unit dose strength of 2 milligram per milliliter (mg/mL).
Drug: Digoxin 0.25 mg — Digoxin will be available as oral tablet at unit dose strength of 0.25 mg.
Drug: Pravastatin 40 mg — Pravastatin will be available as oral tablet at unit dose strength of 40 mg.

SUMMARY:
This is an open-label, single sequence study that is being conducted to investigate the potential drug-drug interaction (DDI) when GSK3640254 is co-administered with a cocktail of cytochrome P450 (CYP) enzymes and transporter probe substrates in healthy participants. This study will aid in understanding these interactions and resulting changes in exposure (if any) when drugs that are metabolized via these pathways are given in combination with GSK3640254. The study will consist of a Screening period and 3 sequential treatment regimens. Participants will be administered a single dose of probe substrate drugs (caffeine 200 milligram (mg), metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg and pravastatin 40 mg) on Day 1. Participants will then receive GSK3640254 200 mg once daily on Days 11 to 20 followed by co-administration of probe substrate drugs with GSK3640254 on Day 21.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination (including cardiopulmonary examination), laboratory tests, and cardiac monitoring (history and ECG).
* Body weight more than or equal to (>=) 50.0 kilograms (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kilogram per square meter (kg/m^2) (inclusive).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants should not engage in intercourse while confined in the clinic. There is no need for an extended period of double barrier use or prolonged abstinence after study discharge.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and at least one of the following conditions applies:
* Is not a woman of childbearing potential (WOCBP) or
* Is a WOCBP and using a non-hormonal contraceptive method that is highly effective, with a failure rate of less than (<) 1 percent (%) for 28 days before intervention, during the intervention period, and for at least 28 days after the last dose of study intervention.
* A WOCBP must have a negative highly sensitive serum pregnancy test at Screening and check-in (Day-1).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions, listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastrointestinal (GI) anatomy or motility (e.g., gastro-esophageal reflux disease, gastric ulcers, gastritis) or hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
* Prior cholecystectomy surgery.
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment.

Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Healthcare (VH)/GlaxoSmithKline (GSK) Medical Monitor.

* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* History of asthma, bronchospasm, or sleep apnea.
* History of chronic musculoskeletal pain (myalgias).
* History of rhabdomyolysis.
* History of a bleeding disorder.
* History of Raynaud's disease.
* History indicative of an increased risk of a cardiac arrhythmia or cardiac disease, including the following:
* History of cardiac arrhythmias or palpitations associated with presyncope or syncope, or history of unexplained syncope.
* History of clinically relevant cardiac disease including symptomatic or asymptomatic arrhythmias (including but not limited to ventricular fibrillation, ventricular tachycardia, any degree of atrioventricular block, Brugada syndrome, Wolff-Parkinson-White syndrome, and sinus bradycardia, defined as heart rate less than 50 beats per minute (bpm) based on vital signs or ECG), presyncope or syncopal episodes, or additional risk factors for torsades de pointes (e.g., heart failure).
* History of clinically relevant structural cardiac disease including hypertrophic obstructive cardiomyopathy.
* History of hypokalemia.
* History of heart disease (e.g., coronary heart disease).
* Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention and positive on reflex to hepatitis C Ribonucleic Acid (RNA).
* Positive HIV-1 and 2 antigen/antibody immunoassay at Screening.
* ALT>=1.5 × upper limit of normal (ULN). A single repeat of ALT is allowed within a single screening period to determine eligibility.
* Bilirubin >=5 × ULN (isolated bilirubin >=5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single screening period to determine eligibility.
* Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT, will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or nonprescription drugs including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Prior exposure to GSK3640254 in another clinical study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia-Suicide Severity Rating Scale (C-SSRS).
* SBP <100 mm Hg. Up to 2 repeats are allowed for confirmation.
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, any degree of atrioventricular block, or conduction abnormality) which will interfere with the safety for the individual participant.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate- <50 or >100 bpm, PR interval- >200 milliseconds and QTcF- >450 milliseconds.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 units. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Unable to refrain from tobacco or nicotine-containing products within 3 months prior to Screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* History of aspirin allergy.
* A participant with known or suspected active coronavirus disease of 2019 (COVID-19) infection OR contact with an individual with known COVID-19, within 14 days of study enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Background] Zhang Y, Johnson M, Joshi S, Yazdani P, Zhan J, Wen B, Bainbridge V, Gartland M, Lataillade M. Open-label, drug-drug interaction study between the HIV-1 maturation inhibitor GSK3640254 and a metabolic probe cocktail in healthy participants. Br J Clin Pharmacol. 2023 Jul;89(7):2236-2245. doi: 10.1111/bcp.15699. Epub 2023 Mar 13. PMID 36822839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States.
Pre-assignment Details: A total of 20 participants were enrolled and received study treatment.
Groups:
- All Treated Participants: All treated participants received a single dose of treatment A: Probe substrates (caffeine 200 milligram [mg], metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) on Day 1; followed by treatment B- GSK3640254 200 mg once daily from Days 11 to 20; further followed by treatment C: Probe substrates (Caffeine 200 mg, metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) co-administered with GSK3640254 200 mg on Day 21.
Period: Treatment Period 1 (Days 1 to 10)
Arm/Group | All Treated Participants
Started | 20
Completed | 20
Not Completed | 0
Period: Treatment Period 2 (Days 11 to 20)
Arm/Group | All Treated Participants
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1
Period: Treatment Period 3 (Days 21 to 26)
Arm/Group | All Treated Participants
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population consisted of all participants who received at least 1 dose of study medication.
Groups:
- All Treated Participants: All treated participants received a single dose of treatment A: Probe substrates (caffeine 200 mg, metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) on Day 1; followed by treatment B- GSK3640254 200 mg once daily from Days 11 to 20; further followed by treatment C: Probe substrates (Caffeine 200 mg, metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) co-administered with GSK3640254 200 mg on Day 21.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.4 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 9
  White - Arabic/North African Heritage | 2
  White - White/Caucasian/European Heritage | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Time t (AUC[0-t]) for Caffeine
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of caffeine. Area under the plasma concentration-time curve from time zero to time t, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, and 120 hours post-dose in treatment period 1 and 3
Population: The Pharmacokinetic (PK) Parameter Population included all participants who underwent plasma PK sampling and had evaluable PK parameters estimated. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter (h*ng/mL)
Groups:
- Treatment A: Probe Substrates: All treated participants received a single dose of treatment A: Probe substrates (caffeine 200 mg, metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) on Day 1.
- Treatment C: Probe Substrates + GSK3640254 200 mg: All treated participants received a single dose of treatment C: Probe substrates (Caffeine 200 mg, metoprolol 100 mg, montelukast 10 mg, flurbiprofen 100 mg, omeprazole 40 mg, midazolam 5 mg, digoxin 0.25 mg, and pravastatin 40 mg) co-administered with GSK3640254 200 mg on Day 21.
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hour*nanograms per milliliter (h*ng/mL) | 37970 (31.1) | 42230 (32.4)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.11, 90% CI 2-sided [0.94 to 1.32] — A mixed-effect model with treatment as a fixed effect and measurements within participant as repeated measures was performed on the natural ln-transformed parameter

2. Primary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC[0-infinity]) for Caffeine
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of caffeine. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 39720 (30.6) | 44440 (30.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.12, 90% CI 2-sided [0.95 to 1.32] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Caffeine
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of caffeine.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Nanograms per milliliter (ng/mL) | 4340 (22.1) | 4110 (25.9)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.95, 90% CI 2-sided [0.83 to 1.08] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Time to Cmax (Tmax) for Caffeine
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of caffeine.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 2.000 [1.00 to 6.00] | 3.000 [0.50 to 6.00]

5. Primary Outcome: Apparent Terminal Phase Half-life (t1/2) for Caffeine
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of caffeine.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 5.380 (21.2) | 6.085 (17.4)

6. Primary Outcome: AUC(0-t) for Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of metoprolol. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 655.0 (135.2) | 807.3 (136.4)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.23, 90% CI 2-sided [0.71 to 2.14] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: AUC(0-infinity) for Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of metoprolol. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 659.1 (134.4) | 813.1 (135.3)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.23, 90% CI 2-sided [0.71 to 2.14] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Cmax for Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of metoprolol.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 127.4 (90.0) | 141.1 (94.4)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.11, 90% CI 2-sided [0.72 to 1.69] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Tmax for Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of metoprolol.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 2.000 [1.00 to 6.00] | 3.000 [1.00 to 4.00]

10. Primary Outcome: t1/2 for Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of metoprolol.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 4.872 (65.6) | 5.342 (59.6)

11. Primary Outcome: AUC(0-t) for Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of montelukast. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 2724 (19.9) | 2940 (18.4)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.08, 90% CI 2-sided [0.97 to 1.20] — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: AUC(0-infinity) for Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of montelukast. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 2859 (20.6) | 3109 (18.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.09, 90% CI 2-sided [0.98 to 1.21] — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Cmax for Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of montelukast.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Nanograms per milliliter (ng/mL) | 379.8 (25.2) | 393.5 (19.5)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.04, 90% CI 2-sided [0.92 to 1.17] — [estimate comment as in outcome 1, analysis 1]

14. Primary Outcome: Tmax for Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of montelukast.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 5.000 [2.00 to 8.03] | 6.000 [3.00 to 8.07]

15. Primary Outcome: t1/2 for Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of montelukast.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 5.035 (10.2) | 5.135 (7.4)

16. Primary Outcome: AUC(0-t) for Flurbiprofen
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of flurbiprofen. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 64930 (28.9) | 66170 (27.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.02, 90% CI 2-sided [0.88 to 1.18] — [estimate comment as in outcome 1, analysis 1]

17. Primary Outcome: AUC(0-infinity) for Flurbiprofen
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of flurbiprofen. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 66700 (28.1) | 68660 (26.7)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.03, 90% CI 2-sided [0.89 to 1.19] — [estimate comment as in outcome 1, analysis 1]

18. Primary Outcome: Cmax for Flurbiprofen
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of flurbiprofen.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 10220 (24.7) | 10710 (19.8)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.05, 90% CI 2-sided [0.93 to 1.18] — [estimate comment as in outcome 1, analysis 1]

19. Primary Outcome: Tmax for Flurbiprofen
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of flurbiprofen.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 3.000 [1.00 to 8.03] | 4.000 [1.00 to 6.07]

20. Primary Outcome: t1/2 for Flurbiprofen
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of flurbiprofen.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 6.123 (31.0) | 6.088 (30.4)

21. Primary Outcome: AUC(0-t) for Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of omeprazole. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 728.1 (114.7) | 817.9 (82.1)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.12, 90% CI 2-sided [0.72 to 1.75] — [estimate comment as in outcome 1, analysis 1]

22. Primary Outcome: AUC(0-infinity) for Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of omeprazole. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 9 | 11
h*ng/mL | 1127 (98.6) | 1093 (75.5)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.97, 90% CI 2-sided [0.54 to 1.73] — [estimate comment as in outcome 1, analysis 1]

23. Primary Outcome: Cmax for Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of omeprazole.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 224.4 (121.6) | 256.6 (72.0)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.14, 90% CI 2-sided [0.73 to 1.78] — [estimate comment as in outcome 1, analysis 1]

24. Primary Outcome: Tmax for Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of omeprazole.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 6.000 [1.50 to 12.07] | 6.000 [1.50 to 12.00]

25. Primary Outcome: t1/2 for Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of omeprazole.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 9 | 11
Hours | 1.439 (32.0) | 1.219 (28.1)

26. Primary Outcome: AUC(0-t) for Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of midazolam. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 67.11 (31.3) | 62.95 (31.0)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.94, 90% CI 2-sided [0.80 to 1.11] — [estimate comment as in outcome 1, analysis 1]

27. Primary Outcome: AUC(0-infinity) for Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of midazolam. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 70.08 (31.4) | 65.46 (31.2)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.93, 90% CI 2-sided [0.79 to 1.10] — [estimate comment as in outcome 1, analysis 1]

28. Primary Outcome: Cmax for Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of midazolam.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 15.44 (39.5) | 13.95 (42.3)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.90, 90% CI 2-sided [0.73 to 1.12] — [estimate comment as in outcome 1, analysis 1]

29. Primary Outcome: Tmax for Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of midazolam.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 1.000 [0.25 to 2.00] | 1.000 [0.25 to 4.00]

30. Primary Outcome: t1/2 for Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of midazolam.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 5.756 (13.2) | 5.222 (20.6)

31. Primary Outcome: AUC(0-t) for Digoxin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of digoxin. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter (h*pg/mL)
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours*picogram per milliliter (h*pg/mL) | 16690 (21.7) | 17840 (26.9)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.07, 90% CI 2-sided [0.94 to 1.22] — [estimate comment as in outcome 1, analysis 1]

32. Primary Outcome: AUC(0-infinity) for Digoxin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of digoxin. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*pg/mL | 19180 (21.5) | 20090 (27.1)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.05, 90% CI 2-sided [0.92 to 1.19] — [estimate comment as in outcome 1, analysis 1]

33. Primary Outcome: Cmax for Digoxin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of digoxin.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter (pg/mL)
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Picogram per milliliter (pg/mL) | 1026 (48.3) | 1282 (56.5)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.25, 90% CI 2-sided [0.96 to 1.63] — [estimate comment as in outcome 1, analysis 1]

34. Primary Outcome: Tmax for Digoxin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of digoxin.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 3.000 [1.50 to 6.00] | 2.000 [1.00 to 4.00]

35. Primary Outcome: t1/2 for Digoxin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of digoxin.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 40.279 (14.3) | 38.784 (12.0)

36. Primary Outcome: AUC(0-t) for Pravastatin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of pravastatin. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 69.92 (63.9) | 51.03 (75.5)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.73, 90% CI 2-sided [0.52 to 1.03] — [estimate comment as in outcome 1, analysis 1]

37. Primary Outcome: AUC(0-infinity) for Pravastatin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of pravastatin. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 16
h*ng/mL | 72.09 (62.9) | 43.70 (47.5)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.61, 90% CI 2-sided [0.45 to 0.82] — [estimate comment as in outcome 1, analysis 1]

38. Primary Outcome: Cmax for Pravastatin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of pravastatin.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 19.45 (79.8) | 15.19 (76.9)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.78, 90% CI 2-sided [0.54 to 1.14] — [estimate comment as in outcome 1, analysis 1]

39. Primary Outcome: Tmax for Pravastatin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of pravastatin.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 1.500 [0.50 to 6.00] | 3.000 [1.00 to 4.00]

40. Primary Outcome: t1/2 for Pravastatin
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of pravastatin.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 16
Hours | 3.189 (43.4) | 3.156 (47.2)

41. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAE was defined as any untoward medical occurrence that, at any dose, results in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement.
Time Frame: Up to Day 26
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B: GSK3640254 200 mg: All treated participants received a single dose of treatment treatment B- GSK3640254 200 mg once daily from Days 11 to 20.
Arm/Group | Treatment A: Probe Substrates | Treatment B: GSK3640254 200 mg | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 20 | 19
Participants
  AEs | 1 | 5 | 5
  SAEs | 0 | 0 | 0

42. Secondary Outcome: Treatment A: Absolute Values of Platelet Count, Leukocyte Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected to analyze the hematology parameters: platelet count, leukocyte count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
10^9 cells per liter
  Baseline (Day -1): Platelet count | 258.6 (59.14)
  Day 10: Platelet count | 265.9 (60.21)
  Baseline (Day -1): Leukocyte count | 5.64 (1.338)
  Day 10: Leukocyte count | 6.30 (1.343)
  Baseline (Day -1): Neutrophils | 3.1504 (1.25074)
  Day 10: Neutrophils | 3.7430 (1.27763)
  Baseline (Day -1): Lymphocytes | 1.8217 (0.39628)
  Day 10: Lymphocytes | 1.8965 (0.33426)
  Baseline (Day -1): Monocytes | 0.4890 (0.15889)
  Day 10: Monocytes | 0.4515 (0.12708)
  Baseline (Day -1): Eosinophils | 0.1461 (0.15067)
  Day 10: Eosinophils | 0.1610 (0.15071)
  Baseline (Day -1): Basophils | 0.0331 (0.01657)
  Day 10: Basophils | 0.0440 (0.01569)

43. Secondary Outcome: Treatment B: Absolute Values of Platelet Count, Leukocyte Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected to analyze the hematology parameters: platelet count, leukocyte count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
10^9 cells per liter
  Baseline (Day 10): Platelet count | 265.9 (60.21)
  Day 20: Platelet count | 261.9 (58.51)
  Baseline (Day 10): Leukocyte count | 6.30 (1.343)
  Day 20: Leukocyte count | 5.79 (1.192)
  Baseline (Day 10): Neutrophils | 3.7430 (1.27763)
  Day 20: Neutrophils | 3.2680 (1.17833)
  Baseline (Day 10): Lymphocytes | 1.8965 (0.33426)
  Day 20: Lymphocytes | 1.8355 (0.52512)
  Baseline (Day 10): Monocytes | 0.4515 (0.12708)
  Day 20: Monocytes | 0.4435 (0.16662)
  Baseline (Day 10): Eosinophils | 0.1610 (0.15071)
  Day 20: Eosinophils | 0.1920 (0.18981)
  Baseline (Day 10): Basophils | 0.0440 (0.01569)
  Day 20: Basophils | 0.0460 (0.02981)

44. Secondary Outcome: Treatment C: Absolute Values of Platelet Count, Leukocyte Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected to analyze the hematology parameters: platelet count, leukocyte count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
10^9 cells per liter
  Baseline (Day 20): Platelet count | 262.3 (60.09)
  Day 22: Platelet count | 249.2 (51.84)
  Day 25: Platelet count | 260.7 (54.96)
  Baseline (Day 20): Leukocyte count | 5.86 (1.184)
  Day 22: Leukocyte count | 5.81 (1.400)
  Day 25: Leukocyte count | 5.98 (1.255)
  Baseline (Day 20): Neutrophils | 3.3179 (1.18871)
  Day 22: Neutrophils | 3.1925 (1.29353)
  Day 25: Neutrophils | 3.4529 (1.16823)
  Baseline (Day 20): Lymphocytes | 1.8437 (0.53820)
  Day 22: Lymphocytes | 1.8787 (0.57389)
  Day 25: Lymphocytes | 1.9280 (0.63546)
  Baseline (Day 20): Monocytes | 0.4505 (0.16811)
  Day 22: Monocytes | 0.4689 (0.14658)
  Day 25: Monocytes | 0.3576 (0.12355)
  Baseline (Day 20): Eosinophils | 0.1953 (0.19443)
  Day 22: Eosinophils | 0.2282 (0.23748)
  Day 25: Eosinophils | 0.1837 (0.20635)
  Baseline (Day 20): Basophils | 0.0474 (0.02997)
  Day 22: Basophils | 0.0380 (0.02395)
  Day 25: Basophils | 0.0408 (0.02134)

45. Secondary Outcome: Treatment A: Absolute Values of Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Proportion of red blood cells in blood
  Baseline (Day -1) | 0.4188 (0.03442)
  Day 10 | 0.4098 (0.03577)

46. Secondary Outcome: Treatment B: Absolute Values of Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Proportion of red blood cells in blood
  Baseline (Day 10) | 0.4098 (0.03577)
  Day 20 | 0.4216 (0.03420)

47. Secondary Outcome: Treatment C: Absolute Values of Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Proportion of red blood cells in blood
  Baseline (Day 20) | 0.4239 (0.03352)
  Day 22 | 0.4022 (0.04433)
  Day 25 | 0.4168 (0.04079)

48. Secondary Outcome: Treatment A: Absolute Values of Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Grams per liter
  Baseline (Day -1) | 141.9 (13.27)
  Day 10 | 137.7 (13.07)

49. Secondary Outcome: Treatment B: Absolute Values of Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Grams per liter
  Baseline (Day 10) | 137.7 (13.07)
  Day 20 | 140.0 (12.22)

50. Secondary Outcome: Treatment C: Absolute Values of Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Grams per liter
  Baseline (Day 20) | 140.6 (12.21)
  Day 22 | 134.7 (15.54)
  Day 25 | 138.3 (13.83)

51. Secondary Outcome: Treatment A: Absolute Values of Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
10^12 cells per liter
  Baseline (Day -1) | 4.836 (0.4125)
  Day 10 | 4.664 (0.4459)

52. Secondary Outcome: Treatment B: Absolute Values of Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
10^12 cells per liter
  Baseline (Day 10) | 4.664 (0.4459)
  Day 20 | 4.746 (0.3994)

53. Secondary Outcome: Treatment C: Absolute Values of Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
10^12 cells per liter
  Baseline (Day 20) | 4.769 (0.3966)
  Day 22 | 4.608 (0.5308)
  Day 25 | 4.756 (0.4718)

54. Secondary Outcome: Treatment A: Absolute Values of Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Femtoliter
  Baseline (Day -1) | 86.71 (3.748)
  Day 10 | 88.02 (3.938)

55. Secondary Outcome: Treatment B: Absolute Values of Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Femtoliter
  Baseline (Day 10) | 88.02 (3.938)
  Day 20 | 88.96 (4.746)

56. Secondary Outcome: Treatment C: Absolute Values of Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Femtoliter
  Baseline (Day 20) | 89.03 (4.865)
  Day 22 | 87.38 (4.217)
  Day 25 | 87.74 (4.045)

57. Secondary Outcome: Treatment A: Absolute Values of Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Picograms
  Baseline (Day -1) | 29.37 (1.546)
  Day 10 | 29.57 (1.667)

58. Secondary Outcome: Treatment B: Absolute Values of Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Picograms
  Baseline (Day 10) | 29.57 (1.667)
  Day 20 | 29.52 (1.602)

59. Secondary Outcome: Treatment C: Absolute Values of Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Picograms
  Baseline (Day 20) | 29.51 (1.645)
  Day 22 | 29.28 (1.670)
  Day 25 | 29.12 (1.626)

60. Secondary Outcome: Treatment A: Absolute Values of Glucose, Carbon Dioxide, Cholesterol, Triglycerides, Anion Gap, Calcium, Chloride, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: glucose, carbon dioxide, cholesterol, triglycerides, anion gap, calcium, chloride, phosphate, potassium, sodium, urea. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Millimoles per liter
  Baseline (Day -1): Glucose | 5.0348 (0.37437)
  Day 10: Glucose | 4.8211 (0.44125)
  Baseline (Day -1): Carbon Dioxide | 104.1 (2.04)
  Day 10: Carbon Dioxide | 25.4 (2.11)
  Baseline (Day -1): Cholesterol | 4.4570 (1.00121)
  Day 10: Cholesterol | 3.8118 (0.85065)
  Baseline (Day -1): Triglycerides | 1.2232 (0.51018)
  Day 10: Triglycerides | 1.1814 (0.82178)
  Baseline (Day -1): Anion Gap | 7.9 (1.80)
  Day 10: Anion Gap | 13.8 (1.71)
  Baseline (Day -1): Calcium | 2.3765 (0.09976)
  Day 10: Calcium | 2.3141 (0.10267)
  Baseline (Day -1): Chloride | 25.8 (2.10)
  Day 10: Chloride | 103.7 (1.81)
  Baseline (Day -1): Phosphate | 1.1075 (0.16734)
  Day 10: Phosphate | 1.1754 (0.16141)
  Baseline (Day -1): Potassium | 4.48 (0.339)
  Day 10: Potassium | 4.43 (0.256)
  Baseline (Day -1): Sodium | 137.7 (2.00)
  Day 10: Sodium | 138.4 (1.93)
  Baseline (Day -1): Urea | 4.8195 (0.78983)
  Day 10: Urea | 5.9458 (1.43309)

61. Secondary Outcome: Treatment B: Absolute Values of Glucose, Carbon Dioxide, Cholesterol, Triglycerides, Anion Gap, Calcium, Chloride, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: glucose, carbon dioxide, cholesterol, triglycerides, anion gap, calcium, chloride, phosphate, potassium, sodium, and urea. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Millimoles per liter
  Baseline (Day 10): Glucose | 4.8211 (0.44125)
  Day 20: Glucose | 4.7378 (0.45996)
  Baseline (Day 10): Carbon Dioxide | 25.4 (2.11)
  Day 20: Carbon Dioxide | 24.9 (2.11)
  Baseline (Day 10): Cholesterol | 3.8118 (0.85065)
  Day 20: Cholesterol | 3.6915 (0.94881)
  Baseline (Day 10): Triglycerides | 1.1814 (0.82178)
  Day 20: Triglycerides | 1.0825 (0.84563)
  Baseline (Day 10): Anion Gap | 13.8 (1.71)
  Day 20: Anion Gap | 14.5 (2.12)
  Baseline (Day 10): Calcium | 2.3141 (0.10267)
  Day 20: Calcium | 2.3141 (0.08825)
  Baseline (Day 10): Chloride | 103.7 (1.81)
  Day 20: Chloride | 103.6 (2.30)
  Baseline (Day 10): Phosphate | 1.1754 (0.16141)
  Day 20: Phosphate | 1.2593 (0.13294)
  Baseline (Day 10): Potassium | 4.43 (0.256)
  Day 20: Potassium | 4.39 (0.383)
  Baseline (Day 10): Sodium | 138.4 (1.93)
  Day 20: Sodium | 138.6 (1.64)
  Baseline (Day 10): Urea | 5.9458 (1.43309)
  Day 20: Urea | 5.6335 (1.72537)

62. Secondary Outcome: Treatment C: Absolute Values of Glucose, Carbon Dioxide, Cholesterol, Triglycerides, Anion Gap, Calcium, Chloride, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: glucose, carbon dioxide, cholesterol, triglycerides, anion gap, calcium, chloride, phosphate, potassium, sodium and urea. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Millimoles per liter
  Baseline (Day 20): Glucose | 4.7184 (0.46406)
  Day 22: Glucose | 4.8060 (0.37890)
  Day 25: Glucose | 4.8703 (0.40699)
  Baseline (Day 20): Carbon Dioxide | 24.9 (2.12)
  Day 22: Carbon Dioxide | 25.4 (1.74)
  Day 25: Carbon Dioxide | 26.2 (1.80)
  Baseline (Day 20): Cholesterol | 3.6898 (0.97478)
  Day 22: Cholesterol | 3.2543 (0.88216)
  Day 25: Cholesterol | 3.3972 (0.89603)
  Baseline (Day 20): Triglycerides | 1.0783 (0.86858)
  Day 22: Triglycerides | 1.0836 (0.78925)
  Day 25: Triglycerides | 1.1074 (0.81372)
  Baseline (Day 20): Anion Gap | 14.6 (2.14)
  Day 22: Anion Gap | 13.9 (1.27)
  Day 25: Anion Gap | 14.5 (1.95)
  Baseline (Day 20): Calcium | 2.3217 (0.08377)
  Day 22: Calcium | 2.2810 (0.10822)
  Day 25: Calcium | 2.3519 (0.09440)
  Baseline (Day 20): Chloride | 103.4 (2.22)
  Day 22: Chloride | 104.8 (2.02)
  Day 25: Chloride | 102.6 (1.86)
  Baseline (Day 20): Phosphate | 1.2661 (0.13297)
  Day 22: Phosphate | 1.1981 (0.14871)
  Day 25: Phosphate | 1.3477 (0.18638)
  Baseline (Day 20): Potassium | 4.38 (0.392)
  Day 22: Potassium | 4.34 (0.347)
  Day 25: Potassium | 4.35 (0.355)
  Baseline (Day 20): Sodium | 138.6 (1.67)
  Day 22: Sodium | 139.8 (1.34)
  Day 25: Sodium | 139.0 (1.67)
  Baseline (Day 20): Urea | 5.7364 (1.70835)
  Day 22: Urea | 4.9078 (1.44100)
  Day 25: Urea | 5.3099 (1.18355)

63. Secondary Outcome: Treatment A: Absolute Values of Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Micromoles per liter
  Baseline (Day -1): Urate | 347.3632 (69.50981)
  Day 10: Urate | 365.5046 (75.74195)
  Baseline (Day -1): Creatinine | 84.9524 (19.89935)
  Day 10: Creatinine | 86.4110 (21.46247)
  Baseline (Day -1): Bilirubin | 9.8325 (3.13227)
  Day 10: Bilirubin | 8.0028 (3.01005)
  Baseline (Day -1): Direct bilirubin | 2.0520 (0.70177)
  Day 10: Direct bilirubin | 1.7015 (0.63856)

64. Secondary Outcome: Treatment B: Absolute Values of Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Micromoles per liter
  Baseline (Day 10): Urate | 365.5046 (75.74195)
  Day 20: Urate | 337.8464 (76.60060)
  Baseline (Day 10): Creatinine | 86.4110 (21.46247)
  Day 20: Creatinine | 90.7868 (22.81174)
  Baseline (Day 10): Bilirubin | 8.0028 (3.01005)
  Day 20: Bilirubin | 8.6184 (3.04856)
  Baseline (Day 10): Direct bilirubin | 1.7015 (0.63856)
  Day 20: Direct bilirubin | 1.8126 (0.64557)

65. Secondary Outcome: Treatment C: Absolute Values of Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Micromoles per liter
  Baseline (Day 20): Urate | 343.1057 (74.89791)
  Day 22: Urate | 303.0349 (71.88291)
  Day 25: Urate | 340.6013 (67.89995)
  Baseline (Day 20): Creatinine | 92.1686 (22.56047)
  Day 22: Creatinine | 87.3764 (22.63812)
  Day 25: Creatinine | 90.5867 (21.29029)
  Baseline (Day 20): Bilirubin | 8.7480 (3.07497)
  Day 22: Bilirubin | 9.8820 (3.24579)
  Day 25: Bilirubin | 9.0360 (3.89534)
  Baseline (Day 20): Direct bilirubin | 1.8450 (0.64634)
  Day 22: Direct bilirubin | 2.0790 (0.60930)
  Day 25: Direct bilirubin | 1.9980 (0.70286)

66. Secondary Outcome: Treatment A: Absolute Values of Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Grams per liter
  Baseline (Day -1): Albumin | 42.9 (2.95)
  Day 10: Albumin | 42.2 (3.14)
  Baseline (Day -1): Globulin | 27.4 (3.14)
  Day 10: Globulin | 25.9 (3.04)
  Baseline (Day -1): Protein | 70.3 (4.52)
  Day 10: Protein | 68.1 (3.77)

67. Secondary Outcome: Treatment B: Absolute Values of Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Grams per liter
  Baseline (Day 10): Albumin | 42.2 (3.14)
  Day 20: Albumin | 41.4 (3.31)
  Baseline (Day 10): Globulin | 25.9 (3.04)
  Day 20: Globulin | 26.8 (3.58)
  Baseline (Day 10): Protein | 68.1 (3.77)
  Day 20: Protein | 68.2 (4.93)

68. Secondary Outcome: Treatment C: Absolute Values of Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Grams per liter
  Baseline (Day 20): Albumin | 41.6 (3.24)
  Day 22: Albumin | 40.5 (3.82)
  Day 25: Albumin | 42.0 (3.04)
  Baseline (Day 20): Globulin | 26.9 (3.65)
  Day 22: Globulin | 25.1 (3.69)
  Day 25: Globulin | 26.6 (3.67)
  Baseline (Day 20): Protein | 68.5 (4.85)
  Day 22: Protein | 65.6 (5.74)
  Day 25: Protein | 68.6 (4.34)

69. Secondary Outcome: Treatment A: Absolute Values of Creatine Kinase, Lactate Dehydrogenase, Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
International units per liter
  Baseline (Day -1): Creatine kinase | 103.7 (79.68)
  Day 10: Creatine kinase | 66.9 (34.67)
  Baseline (Day -1): Lactate dehydrogenase | 131.3 (19.59)
  Day 10: Lactate dehydrogenase | 114.8 (16.87)
  Baseline (Day -1): ALT | 15.6 (7.66)
  Day 10: ALT | 20.1 (14.66)
  Baseline (Day -1): ALP | 62.7 (18.46)
  Day 10: ALP | 60.8 (18.03)
  Baseline (Day -1): AST | 14.6 (3.89)
  Day 10: AST | 15.6 (5.32)
  Baseline (Day -1): Gamma-glutamyl transferase | 19.1 (7.16)
  Day 10: Gamma-glutamyl transferase | 18.9 (8.10)

70. Secondary Outcome: Treatment B: Absolute Values of Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST, and gamma-glutamyl transferase. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
International units per liter
  Baseline (Day 10): Creatine kinase | 66.9 (34.67)
  Day 20: Creatine kinase | 68.9 (47.98)
  Baseline (Day 10): Lactate dehydrogenase | 114.8 (16.87)
  Day 20: Lactate dehydrogenase | 115.9 (17.00)
  Baseline (Day 10): ALT | 20.1 (14.66)
  Day 20: ALT | 20.3 (12.38)
  Baseline (Day 10): ALP | 60.8 (18.03)
  Day 20: ALP | 58.5 (15.56)
  Baseline (Day 10): AST | 15.6 (5.32)
  Day 20: AST | 16.1 (4.80)
  Baseline (Day 10): Gamma-glutamyl transferase | 18.9 (8.10)
  Day 20: Gamma-glutamyl transferase | 18.3 (7.69)

71. Secondary Outcome: Treatment C: Absolute Values of Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST, gamma-glutamyl transferase. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
International units per liter
  Baseline (Day 20): Creatine kinase | 71.3 (48.03)
  Day 22: Creatine kinase | 65.7 (34.56)
  Day 25: Creatine kinase | 63.8 (30.90)
  Baseline (Day 20): Lactate dehydrogenase | 116.6 (17.13)
  Day 22: Lactate dehydrogenase | 120.6 (23.62)
  Day 25: Lactate dehydrogenase | 119.3 (19.18)
  Baseline (Day 20): ALT | 20.4 (12.70)
  Day 22: ALT | 17.3 (9.36)
  Day 25: ALT | 20.9 (11.92)
  Baseline (Day 20): ALP | 58.5 (15.98)
  Day 22: ALP | 57.6 (16.26)
  Day 25:ALP | 58.6 (16.40)
  Baseline (Day 20): AST | 16.2 (4.91)
  Day 22: AST | 14.7 (3.78)
  Day 25: AST | 16.4 (4.56)
  Baseline (Day 20): Gamma-glutamyl transferase | 18.5 (7.83)
  Day 22: Gamma-glutamyl transferase | 17.1 (6.77)
  Day 25: Gamma-glutamyl transferase | 18.7 (8.23)

72. Secondary Outcome: Treatment A: Absolute Values of Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Units per liter
  Baseline (Day -1): Lipase | 29.4 (14.73)
  Day 10: Lipase | 31.6 (11.99)
  Baseline (Day -1): Amylase | 59.5 (22.37)
  Day 10: Amylase | 56.9 (20.93)

73. Secondary Outcome: Treatment B: Absolute Values of Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Units per liter
  Baseline (Day 10): Lipase | 31.6 (11.99)
  Day 20: Lipase | 32.4 (14.51)
  Baseline (Day 10): Amylase | 56.9 (20.93)
  Day 20: Amylase | 60.1 (23.22)

74. Secondary Outcome: Treatment C: Absolute Values of Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Units per liter
  Baseline (Day 20): Lipase | 32.9 (14.74)
  Day 22: Lipase | 33.5 (15.19)
  Day 25: Lipase | 33.1 (14.58)
  Baseline (Day 20): Amylase | 62.2 (21.79)
  Day 22: Amylase | 64.7 (25.32)
  Day 25: Amylase | 60.7 (21.08)

75. Secondary Outcome: Treatment A: Change From Baseline in Platelet Count, Leukocyte Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected to analyze the hematology parameters: platelet count, leukocyte count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
10^9 cells per liter
  Platelet count | 7.3 (20.01)
  Leukocyte count | 0.66 (0.844)
  Neutrophils | 0.5926 (0.68577)
  Lymphocytes | 0.0748 (0.25872)
  Monocytes | -0.0375 (0.09379)
  Eosinophils | 0.0150 (0.07023)
  Basophils | 0.0110 (0.02138)

76. Secondary Outcome: Treatment B: Change From Baseline in Platelet Count, Leukocyte Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected to analyze the hematology parameters: platelet count, leukocyte count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
10^9 cells per liter
  Platelet count | -4.1 (17.31)
  Leukocyte count | -0.51 (0.947)
  Neutrophils | -0.4750 (0.63752)
  Lymphocytes | -0.0610 (0.39045)
  Monocytes | -0.0080 (0.11134)
  Eosinophils | 0.0310 (0.10686)
  Basophils | 0.0020 (0.02526)

77. Secondary Outcome: Treatment C: Change From Baseline in Platelet Count, Leukocyte Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected to analyze the hematology parameters: platelet count, leukocyte count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
10^9 cells per liter
  Day 22: Platelet count | -13.1 (19.31)
  Day 25: Platelet count | -1.6 (24.62)
  Day 22: Leukocyte count | -0.05 (0.906)
  Day 25: Leukocyte count | 0.12 (0.820)
  Day 22: Neutrophils | -0.1254 (0.74916)
  Day 25: Neutrophils | 0.1351 (0.72701)
  Day 22: Lymphocytes | 0.0351 (0.42962)
  Day 25: Lymphocytes | 0.0843 (0.41536)
  Day 22: Monocytes | 0.0184 (0.08808)
  Day 25: Monocytes | -0.0929 (0.17694)
  Day 22: Eosinophils | 0.0329 (0.12007)
  Day 25: Eosinophils | -0.0115 (0.06076)
  Day 22: Basophils | -0.0094 (0.03787)
  Day 25: Basophils | -0.0066 (0.03173)

78. Secondary Outcome: Treatment A: Change From Baseline in Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Proportion of red blood cells in blood | -0.0090 (0.02082)

79. Secondary Outcome: Treatment B: Change From Baseline in Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Proportion of red blood cells in blood | 0.0118 (0.01667)

80. Secondary Outcome: Treatment C: Change From Baseline in Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Proportion of red blood cells in blood
  Day 22 | -0.0217 (0.02090)
  Day 25 | -0.0071 (0.02129)

81. Secondary Outcome: Treatment A: Change From Baseline in Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Grams per liter | -4.2 (6.34)

82. Secondary Outcome: Treatment B: Change From Baseline in Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Grams per liter | 2.3 (4.91)

83. Secondary Outcome: Treatment C: Change From Baseline in Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Grams per liter
  Day 22 | -5.8 (6.52)
  Day 25 | -2.3 (5.82)

84. Secondary Outcome: Treatment A: Change From Baseline in Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
10^12 cells per liter | -0.172 (0.2219)

85. Secondary Outcome: Treatment B: Change From Baseline in Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
10^12 cells per liter | 0.083 (0.1768)

86. Secondary Outcome: Treatment C: Change From Baseline in Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
10^12 cells per liter
  Day 22 | -0.161 (0.2190)
  Day 25 | -0.013 (0.2027)

87. Secondary Outcome: Treatment A: Change From Baseline in Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Femtoliter | 1.31 (1.539)

88. Secondary Outcome: Treatment B: Change From Baseline in Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Femtoliter | 0.94 (2.519)

89. Secondary Outcome: Treatment C: Change From Baseline in Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Femtoliter
  Day 22 | -1.64 (1.849)
  Day 25 | -1.28 (2.234)

90. Secondary Outcome: Treatment A: Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Picograms | 0.20 (0.352)

91. Secondary Outcome: Treatment B: Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Picograms | -0.05 (0.298)

92. Secondary Outcome: Treatment C: Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Picograms
  Day 22 | -0.23 (0.407)
  Day 25 | -0.39 (0.519)

93. Secondary Outcome: Treatment A: Change From Baseline in Glucose, Carbon Dioxide, Cholesterol, Triglycerides, Anion Gap, Calcium, Chloride, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: glucose, carbon dioxide, cholesterol, triglycerides, anion gap, calcium, chloride, phosphate, potassium, sodium, and urea. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Millimoles per liter
  Glucose | -0.2137 (0.29663)
  Carbon Dioxide | -78.7 (3.12)
  Cholesterol | -0.6452 (0.47501)
  Triglycerides | -0.0418 (0.59458)
  Anion Gap | 5.9 (2.21)
  Calcium | -0.0624 (0.04889)
  Chloride | 78.0 (2.98)
  Phosphate | 0.0678 (0.10522)
  Potassium | -0.05 (0.402)
  Sodium | 0.7 (2.16)
  Urea | 1.1263 (0.97483)

94. Secondary Outcome: Treatment B: Change From Baseline in Glucose, Carbon Dioxide, Cholesterol, Triglycerides, Anion Gap, Calcium, Chloride, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: glucose, carbon dioxide, cholesterol, triglycerides, anion gap, calcium, chloride, phosphate, potassium, sodium, and urea. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Millimoles per liter
  Glucose | -0.0833 (0.29345)
  Carbon Dioxide | -0.6 (1.79)
  Cholesterol | -0.1203 (0.30774)
  Triglycerides | -0.0989 (0.30531)
  Anion Gap | 0.8 (1.94)
  Calcium | 0.0000 (0.06575)
  Chloride | -0.1 (1.52)
  Phosphate | 0.0840 (0.08601)
  Potassium | -0.05 (0.378)
  Sodium | 0.3 (1.41)
  Urea | -0.3124 (0.72202)

95. Secondary Outcome: Treatment C: Change From Baseline in Glucose, Carbon Dioxide, Cholesterol, Triglycerides, Anion Gap, Calcium, Chloride, Phosphate, Potassium, Sodium, Urea
Description: Blood samples were collected to analyze the chemistry parameters: glucose, carbon dioxide, cholesterol, triglycerides, anion gap, calcium, chloride, phosphate, potassium, sodium and urea. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Millimoles per liter
  Day 22: Glucose | 0.0876 (0.29392)
  Day 25: Glucose | 0.1519 (0.32570)
  Day 22: Carbon Dioxide | 0.5 (2.12)
  Day 25: Carbon Dioxide | 1.2 (1.81)
  Day 22: Cholesterol | -0.4355 (0.31287)
  Day 25: Cholesterol | -0.2926 (0.25147)
  Day 22: Triglycerides | 0.0054 (0.14595)
  Day 25: Triglycerides | 0.0291 (0.18280)
  Day 22: Anion Gap | -0.6 (1.80)
  Day 25: Anion Gap | -0.1 (0.97)
  Day 22: Calcium | -0.0407 (0.07165)
  Day 25: Calcium | 0.0302 (0.05553)
  Day 22: Chloride | 1.4 (1.64)
  Day 25: Chloride | -0.8 (1.78)
  Day 22: Phosphate | -0.0680 (0.09860)
  Day 25: Phosphate | 0.0816 (0.09527)
  Day 22: Potassium | -0.04 (0.373)
  Day 25: Potassium | -0.03 (0.441)
  Day 22: Sodium | 1.2 (1.51)
  Day 25: Sodium | 0.4 (2.41)
  Day 22: Urea | -0.8286 (0.88169)
  Day 25: Urea | -0.4265 (0.85981)

96. Secondary Outcome: Treatment A: Change From Baseline in Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Micromoles per liter
  Urate | 18.1414 (39.28786)
  Creatinine | 1.4586 (5.65145)
  Bilirubin | -1.8297 (1.38266)
  Direct bilirubin | -0.3506 (0.60895)

97. Secondary Outcome: Treatment B: Change From Baseline in Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Micromoles per liter
  Urate | -27.6582 (25.47573)
  Creatinine | 4.3758 (4.38239)
  Bilirubin | 0.6156 (1.92059)
  Direct bilirubin | 0.1112 (0.46509)

98. Secondary Outcome: Treatment C: Change From Baseline in Urate, Creatinine, Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: urate, creatinine, bilirubin and direct bilirubin. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Micromoles per liter
  Day 22: Urate | -40.0707 (26.51457)
  Day 25: Urate | -2.5044 (26.62359)
  Day 22: Creatinine | -4.7922 (5.82901)
  Day 25: Creatinine | -1.5819 (4.60830)
  Day 22: Bilirubin | 1.1340 (1.91202)
  Day 25: Bilirubin | 0.2880 (2.14494)
  Day 22: Direct bilirubin | 0.2340 (0.38326)
  Day 25: Direct bilirubin | 0.1530 (0.39447)

99. Secondary Outcome: Treatment A: Change From Baseline in Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Grams per liter
  Albumin | -0.7 (1.75)
  Globulin | -1.5 (1.61)
  Protein | -2.2 (2.57)

100. Secondary Outcome: Treatment B: Change From Baseline in Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Grams per liter
  Albumin | -0.9 (2.43)
  Globulin | 0.9 (2.07)
  Protein | 0.1 (3.71)

101. Secondary Outcome: Treatment C: Change From Baseline in Albumin, Globulin, Protein
Description: Blood samples were collected to analyze the chemistry parameters: albumin, globulin and protein. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Grams per liter
  Day 22: Albumin | -1.1 (2.44)
  Day 25: Albumin | 0.4 (1.71)
  Day 22: Globulin | -1.8 (1.98)
  Day 25: Globulin | -0.3 (1.76)
  Day 22: Protein | -2.9 (4.15)
  Day 25: Protein | 0.2 (2.81)

102. Secondary Outcome: Treatment A: Change From Baseline in Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST and gamma-glutamyl transferase. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
International units per liter
  Creatine kinase | -36.9 (59.38)
  Lactate dehydrogenase | -16.5 (15.50)
  ALT | 4.5 (11.51)
  ALP | -1.9 (6.39)
  AST | 1.0 (4.52)
  Gamma-glutamyl transferase | -0.2 (3.86)

103. Secondary Outcome: Treatment B: Change From Baseline in Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST, and gamma-glutamyl transferase. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
International units per liter
  Creatine kinase | 2.1 (24.48)
  Lactate dehydrogenase | 1.1 (13.15)
  ALT | 0.3 (6.78)
  ALP | -2.4 (6.21)
  AST | 0.6 (3.03)
  Gamma-glutamyl transferase | -0.6 (2.74)

104. Secondary Outcome: Treatment C: Change From Baseline in Creatine Kinase, Lactate Dehydrogenase, ALT, ALP, AST, Gamma-glutamyl Transferase
Description: Blood samples were collected to analyze the chemistry parameters: creatine kinase, lactate dehydrogenase, ALT, ALP, AST, gamma-glutamyl transferase. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
International units per liter
  Day 22: Creatine kinase | -5.6 (21.78)
  Day 25: Creatine kinase | -7.5 (26.10)
  Day 22: Lactate dehydrogenase | 4.0 (18.94)
  Day 25: Lactate dehydrogenase | 2.6 (16.30)
  Day 22: ALT | -3.1 (4.12)
  Day 25: ALT | 0.5 (2.61)
  Day 22: ALP | -0.9 (5.83)
  Day 25:ALP | 0.1 (3.91)
  Day 22: AST | -1.5 (2.78)
  Day 25: AST | 0.2 (1.89)
  Day 22: Gamma-glutamyl transferase | -1.5 (1.61)
  Day 25: Gamma-glutamyl transferase | 0.2 (1.26)

105. Secondary Outcome: Treatment A: Change From Baseline in Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day -1), before the dose of Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day -1) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Units per liter
  Lipase | 2.2 (6.81)
  Amylase | -2.6 (7.86)

106. Secondary Outcome: Treatment B: Change From Baseline in Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 10), before the first dose of Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 10) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Units per liter
  Lipase | 0.9 (6.07)
  Amylase | 3.2 (6.31)

107. Secondary Outcome: Treatment C: Change From Baseline in Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 20), before the dose of Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 20), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Units per liter
  Day 22: Lipase | 0.6 (10.08)
  Day 25: Lipase | 0.2 (4.88)
  Day 22: Amylase | 2.5 (7.10)
  Day 25: Amylase | -1.5 (4.98)

108. Secondary Outcome: Treatment A: Absolute Values for Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Fridericia's Formula (QTcF)
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A.
Time Frame: Baseline (Day 1, Pre-Dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Milliseconds
  Baseline (Day 1, Pre-dose): PR Interval | 154.8 (20.92)
  Day 10: PR Interval | 158.2 (22.67)
  Baseline (Day 1, Pre-dose): QRS Duration | 92.5 (8.34)
  Day 10: QRS Duration | 95.0 (10.11)
  Baseline (Day 1, Pre-dose): QT Interval | 391.2 (22.41)
  Day 10: QT Interval | 398.3 (22.19)
  Baseline (Day 1, Pre-dose): QTcF Interval | 401.0 (16.48)
  Day 10: QTcF Interval | 405.8 (16.25)

109. Secondary Outcome: Treatment B: Absolute Values for ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF Interval
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Milliseconds
  Baseline (Day 11, Pre-dose): PR Interval | 158.6 (19.44)
  Day 20: PR Interval | 161.8 (22.40)
  Baseline (Day 11, Pre-dose): QRS Duration | 94.2 (8.73)
  Day 20: QRS Duration | 96.4 (9.25)
  Baseline (Day 11, Pre-dose): QT Interval | 403.1 (26.27)
  Day 20: QT Interval | 408.8 (25.85)
  Baseline (Day 11, Pre-dose): QTcF Interval | 403.5 (17.63)
  Day 20: QTcF Interval | 408.6 (17.26)

110. Secondary Outcome: Treatment C: Absolute Values for ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF Interval
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Milliseconds
  Baseline (Day 21, Pre-dose): PR Interval | 160.8 (20.26)
  Day 22: PR Interval | 162.3 (22.07)
  Day 25: PR Interval | 159.6 (23.55)
  Baseline (Day 21, Pre-dose): QRS Duration | 95.8 (9.49)
  Day 22: QRS Duration | 98.7 (10.30)
  Day 25: QRS Duration | 96.8 (8.42)
  Baseline (Day 21, Pre-dose): QT Interval | 402.6 (21.06)
  Day 22: QT Interval | 420.6 (21.16)
  Day 25: QT Interval | 398.7 (22.25)
  Baseline (Day 21, Pre-dose): QTcF Interval | 408.7 (16.31)
  Day 22: QTcF Interval | 407.3 (13.75)
  Day 25: QTcF Interval | 402.5 (17.03)

111. Secondary Outcome: Treatment A: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Milliseconds
  PR Interval | 3.4 (9.28)
  QRS Duration | 2.5 (4.37)
  QT Interval | 7.1 (12.81)
  QTcF Interval | 4.8 (9.27)

112. Secondary Outcome: Treatment B: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Milliseconds
  PR Interval | 3.2 (8.79)
  QRS Duration | 2.3 (2.77)
  QT Interval | 5.7 (13.30)
  QTcF Interval | 5.1 (10.69)

113. Secondary Outcome: Treatment C: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcF
Description: Twelve-lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Milliseconds
  Day 22: PR Interval | 1.5 (9.99)
  Day 25: PR Interval | -1.2 (10.07)
  Day 22: QRS Duration | 2.9 (4.24)
  Day 25: QRS Duration | 1.0 (3.43)
  Day 22: QT Interval | 18.0 (20.32)
  Day 25: QT Interval | -3.9 (16.18)
  Day 22: QTcF Interval | -1.4 (9.44)
  Day 25: QTcF Interval | -6.3 (8.41)

114. Secondary Outcome: Treatment A: Absolute Values of Oral Temperature
Description: Oral temperature was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Degrees Celsius
  Baseline (Day 1, Pre-dose) | 36.38 (0.293)
  Day 10 | 36.26 (0.252)

115. Secondary Outcome: Treatment B: Absolute Values of Oral Temperature
Description: Oral temperature was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Degrees Celsius
  Baseline (Day 11, Pre-dose) | 36.31 (0.320)
  Day 20 | 36.28 (0.246)

116. Secondary Outcome: Treatment C: Absolute Values of Oral Temperature
Description: Oral temperature was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Degrees Celsius
  Baseline (Day 21, Pre-dose) | 36.31 (0.284)
  Day 22 | 36.18 (0.210)
  Day 25 | 36.31 (0.300)

117. Secondary Outcome: Treatment A: Absolute Values of Pulse Rate
Description: Pulse rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Beats per minute
  Baseline (Day 1, Pre-dose) | 64.5 (8.97)
  Day 10 | 65.0 (8.19)

118. Secondary Outcome: Treatment B: Absolute Values of Pulse Rate
Description: Pulse rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Beats per minute
  Baseline (Day 11, Pre-dose) | 61.6 (9.95)
  Day 20 | 62.8 (10.22)

119. Secondary Outcome: Treatment C: Absolute Values of Pulse Rate
Description: Pulse rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Beats per minute
  Baseline (Day 21, Pre-dose) | 63.2 (7.04)
  Day 22 | 56.2 (6.83)
  Day 25 | 61.7 (7.27)

120. Secondary Outcome: Treatment A: Absolute Values of Respiratory Rate
Description: Respiratory rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A.
Time Frame: Baseline (Day 1, Pre-dose) and Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Breaths per minute
  Baseline (Day 1, Pre-dose) | 16.1 (1.37)
  Day 2 | 15.8 (2.33)

121. Secondary Outcome: Treatment B: Absolute Values of Respiratory Rate
Description: Respiratory rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Breaths per minute
  Baseline (Day 11, Pre-dose) | 15.0 (2.29)
  Day 20 | 14.7 (2.27)

122. Secondary Outcome: Treatment C: Absolute Values of Respiratory Rate
Description: Respiratory rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Breaths per minute
  Baseline (Day 21, Pre-dose) | 15.7 (1.56)
  Day 22 | 15.7 (1.38)
  Day 25 | 16.5 (2.20)

123. Secondary Outcome: Treatment A: Absolute Values of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Millimeters of mercury
  Baseline (Day 1, Pre-dose): SBP | 111.0 (9.03)
  Day 10: SBP | 107.7 (9.32)
  Baseline (Day 1, Pre-dose): DBP | 65.1 (6.73)
  Day 10: DBP | 59.7 (6.24)

124. Secondary Outcome: Treatment B: Absolute Values of SBP and DBP
Description: SBP and DBP were measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Millimeters of mercury
  Baseline (Day 11, Pre-dose): SBP | 107.7 (8.46)
  Day 20: SBP | 107.2 (9.52)
  Baseline (Day 11, Pre-dose): DBP | 61.6 (6.56)
  Day 20: DBP | 59.6 (5.55)

125. Secondary Outcome: Treatment C: Absolute Values of SBP and DBP
Description: SBP and DBP were measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Millimeters of mercury
  Baseline (Day 21, Pre-dose): SBP | 107.5 (8.49)
  Day 22: SBP | 105.6 (11.93)
  Day 25: SBP | 109.7 (7.96)
  Baseline (Day 21, Pre-dose): DBP | 62.7 (5.31)
  Day 22: DBP | 58.4 (5.87)
  Day 25: DBP | 62.2 (5.06)

126. Secondary Outcome: Treatment A: Change From Baseline in Oral Temperature
Description: Oral temperature was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Degrees Celsius | -0.12 (0.314)

127. Secondary Outcome: Treatment B: Change From Baseline in Oral Temperature
Description: Oral temperature was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Degrees Celsius | -0.03 (0.249)

128. Secondary Outcome: Treatment C: Change From Baseline in Oral Temperature
Description: Oral temperature was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Degrees Celsius
  Day 22 | -0.13 (0.242)
  Day 25 | 0.01 (0.286)

129. Secondary Outcome: Treatment A: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Beats per minute | 0.5 (6.27)

130. Secondary Outcome: Treatment B: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Beats per minute | 1.3 (7.44)

131. Secondary Outcome: Treatment C: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Beats per minute
  Day 22 | -7.1 (7.48)
  Day 25 | -1.5 (6.17)

132. Secondary Outcome: Treatment A: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Breaths per minute | -0.3 (2.62)

133. Secondary Outcome: Treatment B: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Breaths per minute | -0.3 (2.36)

134. Secondary Outcome: Treatment C: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Breaths per minute
  Day 22 | -0.1 (1.90)
  Day 25 | 0.8 (2.37)

135. Secondary Outcome: Treatment A: Change From Baseline in SBP and DBP
Description: SBP and DBP were measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment A was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 1, Pre-Dose), before the dose in Treatment A. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1, Pre-dose) and Day 10
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment A: Probe Substrates
Number analyzed (Participants) | 20
Millimeters of mercury
  SBP | -3.3 (9.67)
  DBP | -5.4 (5.96)

136. Secondary Outcome: Treatment B: Change From Baseline in SBP and DBP
Description: SBP and DBP were measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment B was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 11, Pre-Dose), before the first dose in Treatment B. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 11, Pre-Dose) and Day 20
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment B: GSK3640254 200 mg
Number analyzed (Participants) | 20
Millimeters of mercury
  SBP | -0.5 (8.56)
  DBP | -2.0 (5.75)

137. Secondary Outcome: Treatment C: Change From Baseline in SBP and DBP
Description: SBP and DBP were measured in the supine position after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline for treatment C was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits (Day 21, Pre-Dose), before the first dose in Treatment C. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 21, Pre-Dose), Days 22 and 25
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Millimeters of mercury
  Day 22: SBP | -1.9 (10.84)
  Day 25: SBP | 2.2 (8.67)
  Day 22: DBP | -4.3 (4.75)
  Day 25: DBP | -0.5 (4.78)

138. Secondary Outcome: Treatment C: AUC(0-t) for GSK3640254
Description: Blood samples were collected at the indicated time points for steady-state pharmacokinetic analysis of GSK3640254. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: Pre-dose and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72, 96, and 120 hours post-dose in treatment period 3
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
h*ng/mL | 51840 (48.8)

139. Secondary Outcome: Treatment C: AUC From Time Zero to the End of the Dosing Interval at Steady State (AUC[0-tau]) for GSK3640254
Description: Blood samples were collected at the indicated time points for steady-state pharmacokinetic analysis of GSK3640254.
Time Frame: as for outcome 138
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
h*ng/mL | 22920 (37.3)

140. Secondary Outcome: Treatment C: Cmax for GSK3640254
Description: Blood samples were collected at the indicated time points for steady-state pharmacokinetic analysis of GSK3640254.
Time Frame: as for outcome 138
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
ng/mL | 1450 (41.7)

141. Secondary Outcome: Treatment C: Plasma Concentration at the End of the Dosing Interval (Ctau) for GSK3640254
Description: Blood samples were collected at the indicated time points for steady-state pharmacokinetic analysis of GSK3640254.
Time Frame: as for outcome 138
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
ng/mL | 729.5 (35.5)

142. Secondary Outcome: Treatment C: Tmax for GSK3640254
Description: Blood samples were collected at the indicated time points for steady-state pharmacokinetic analysis of GSK3640254.
Time Frame: as for outcome 138
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19
Hours | 4.500 [2.00 to 8.03]

143. Secondary Outcome: Treatment C: t1/2 for GSK3640254
Description: Blood samples were collected at the indicated time points for steady-state pharmacokinetic analysis of GSK3640254.
Time Frame: as for outcome 138
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 18
Hours | 29.556 (16.9)

144. Secondary Outcome: AUC(0-t) for Alpha-hydroxymetoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of alpha-hydroxymetoprolol. Alpha-hydroxymetoprolol is a metabolite of metoprolol. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 531.3 (159.4) | 487.9 (174.4)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.92, 90% CI 2-sided [0.49 to 1.71] — [estimate comment as in outcome 1, analysis 1]

145. Secondary Outcome: AUC(0-infinity) for Alpha-hydroxymetoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of alpha-hydroxymetoprolol. Alpha-hydroxymetoprolol is a metabolite of metoprolol. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19 | 18
h*ng/mL | 682.8 (34.1) | 632.8 (50.7)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.93, 90% CI 2-sided [0.74 to 1.16] — [estimate comment as in outcome 1, analysis 1]

146. Secondary Outcome: Cmax for Alpha-hydroxymetoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of alpha-hydroxymetoprolol. Alpha-hydroxymetoprolol is a metabolite of metoprolol.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 45.70 (199.8) | 39.21 (212.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.86, 90% CI 2-sided [0.43 to 1.72] — [estimate comment as in outcome 1, analysis 1]

147. Secondary Outcome: Tmax for Alpha-hydroxymetoprolol
Description: as for outcome 146
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 3.033 [1.00 to 6.00] | 4.000 [1.00 to 8.00]

148. Secondary Outcome: t1/2 for Alpha-hydroxymetoprolol
Description: as for outcome 146
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 19 | 18
Hours | 8.040 (31.4) | 8.339 (23.0)

149. Secondary Outcome: AUC(0-t) for 36-hydroxymontelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 36-hydroxymontelukas. 36-hydroxymontelukast is a metabolite of montelukast. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 234.2 (47.2) | 230.9 (59.1)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.99, 90% CI 2-sided [0.75 to 1.29] — [estimate comment as in outcome 1, analysis 1]

150. Secondary Outcome: AUC(0-infinity) for 36-hydroxymontelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 36-hydroxymontelukast. 36-hydroxymontelukast is a metabolite of montelukast. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 252.5 (48.2) | 249.3 (58.7)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.99, 90% CI 2-sided [0.75 to 1.29] — [estimate comment as in outcome 1, analysis 1]

151. Secondary Outcome: Cmax for 36-hydroxymontelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 36-hydroxymontelukast. 36-hydroxymontelukast is a metabolite of montelukast.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 24.62 (45.7) | 23.22 (55.0)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.94, 90% CI 2-sided [0.73 to 1.22] — [estimate comment as in outcome 1, analysis 1]

152. Secondary Outcome: Tmax for 36-hydroxymontelukast
Description: as for outcome 151
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 6.000 [3.00 to 8.03] | 6.000 [4.00 to 8.13]

153. Secondary Outcome: t1/2 for 36-hydroxymontelukast
Description: as for outcome 151
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 5.310 (14.3) | 5.644 (15.1)

154. Secondary Outcome: AUC(0-t) for 5-hydroxyomeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 5-hydroxyomeprazole. 5-hydroxyomeprazole is a metabolite of omeprazole. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 713.5 (38.0) | 785.1 (24.7)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.10, 90% CI 2-sided [0.93 to 1.30] — [estimate comment as in outcome 1, analysis 1]

155. Secondary Outcome: AUC(0-infinity) for 5-hydroxyomeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 5-hydroxyomeprazole. 5-hydroxyomeprazole is a metabolite of omeprazole. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 14 | 14
h*ng/mL | 767.4 (30.9) | 762.0 (25.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.99, 90% CI 2-sided [0.83 to 1.19] — [estimate comment as in outcome 1, analysis 1]

156. Secondary Outcome: Cmax for 5-hydroxyomeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 5-hydroxyomeprazole. 5-hydroxyomeprazole is a metabolite of omeprazole.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 181.1 (63.1) | 203.3 (28.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 1.12, 90% CI 2-sided [0.88 to 1.44] — [estimate comment as in outcome 1, analysis 1]

157. Secondary Outcome: Tmax for 5-hydroxyomeprazole
Description: as for outcome 156
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 6.000 [2.05 to 12.07] | 6.000 [1.50 to 12.00]

158. Secondary Outcome: t1/2 for 5-hydroxyomeprazole
Description: as for outcome 156
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 14 | 14
Hours | 1.580 (15.4) | 1.569 (13.5)

159. Secondary Outcome: AUC(0-t) for 1-hydroxymidazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 1-hydroxymidazolam. 1-hydroxymidazolam is a metabolite of midazolam. The AUC(0-t) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 31.07 (33.0) | 28.07 (37.0)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.90, 90% CI 2-sided [0.75 to 1.09] — [estimate comment as in outcome 1, analysis 1]

160. Secondary Outcome: AUC(0-infinity) for 1-hydroxymidazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 1-hydroxymidazolam. 1-hydroxymidazolam is a metabolite of midazolam. The AUC(0-infinity) was determined using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
h*ng/mL | 31.86 (32.5) | 28.99 (36.6)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.91, 90% CI 2-sided [0.76 to 1.09] — [estimate comment as in outcome 1, analysis 1]

161. Secondary Outcome: Cmax for 1-hydroxymidazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of 1-hydroxymidazolam. 1-hydroxymidazolam is a metabolite of midazolam.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
ng/mL | 7.933 (53.8) | 6.722 (48.1)
Statistical Analysis 1: Comparison: Treatment A: Probe Substrates vs Treatment C: Probe Substrates + GSK3640254 200 mg; Test type: Other; Ratio of geometric least square mean = 0.85, 90% CI 2-sided [0.65 to 1.10] — [estimate comment as in outcome 1, analysis 1]

162. Secondary Outcome: Tmax for 1-hydroxymidazolam
Description: as for outcome 161
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 1.000 [0.25 to 3.00] | 1.000 [0.25 to 4.00]

163. Secondary Outcome: t1/2 for 1-hydroxymidazolam
Description: as for outcome 161
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Hours | 3.632 (15.6) | 3.717 (21.0)

164. Secondary Outcome: Ratio of Cmax of Alpha-hydroxymetoprolol to Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (metoprolol) and its metabolite (alpha-hydroxymetoprolol). Ratio of Cmax of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 0.7869 (0.76896) | 0.7066 (0.93732)

165. Secondary Outcome: Ratio of AUC(0-infinity) of Alpha-hydroxymetoprolol to Metoprolol
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (metoprolol) and its metabolite (alpha-hydroxymetoprolol). Ratio of AUC(0-infinity) of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 1.733 (1.6208) | 1.449 (1.6511)

166. Secondary Outcome: Ratio of Cmax of 36-hydroxymontelukast to Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (montelukast) and its metabolite (36-hydroxymontelukast). Ratio of Cmax of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 0.06766 (0.025068) | 0.06308 (0.025951)

167. Secondary Outcome: Ratio of AUC(0-infinity) of 36-hydroxymontelukast to Montelukast
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (montelukast) and its metabolite (36-hydroxymontelukast). Ratio of AUC(0-infinity) of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 0.09182 (0.033472) | 0.08562 (0.036555)

168. Secondary Outcome: Ratio of Cmax of 5-hydroxyomeprazole to Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (omeprazole) and its metabolite (5-hydroxyomeprazole). Ratio of Cmax of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 0.9461 (0.56833) | 0.8810 (0.49954)

169. Secondary Outcome: Ratio of AUC(0-infinity) of 5-hydroxyomeprazole to Omeprazole
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (omeprazole) and its metabolite (5-hydroxyomeprazole). Ratio of AUC(0-infinity) of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 1.151 (0.66463) | 1.077 (0.59178)

170. Secondary Outcome: Ratio of Cmax of 1-hydroxymidazolam to Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (midazolam) and its metabolite (1-hydroxymidazolam). Ratio of Cmax of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 0.5286 (0.23819) | 0.4955 (0.20616)

171. Secondary Outcome: Ratio of AUC(0-infinity) of 1-hydroxymidazolam to Midazolam
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of parent drug (midazolam) and its metabolite (1-hydroxymidazolam). Ratio of AUC(0-infinity) of metabolite to parent drug has been presented.
Time Frame: as for outcome 1
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment A: Probe Substrates | Treatment C: Probe Substrates + GSK3640254 200 mg
Number analyzed (Participants) | 20 | 19
Ratio | 0.4677 (0.19853) | 0.4618 (0.20637)

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to Day 26
Description: Safety Population consisted of all participants who received at least 1 dose of study medication.
Arm/Group | Treatment A: Probe Substrates | Treatment B: GSK3640254 200 mg | Treatment C: Probe Substrates + GSK3640254 200 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/20 | 5/20 | 5/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Probe Substrates (N=20) | Treatment B: GSK3640254 200 mg (N=20) | Treatment C: Probe Substrates + GSK3640254 200 mg (N=19)
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT04425902/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT04425902/SAP_001.pdf